CLINICAL TRIAL: NCT06473480
Title: Continuous GLUCOse Monitoring System With a SENSor Compared to Fingerstick Glucose Monitoring in Surgical Wards (GLUCOSENS)
Brief Title: Continuous Bloodsugar Monitoring System With a Sensor Compared to Fingerstick Bloodsugar Monitoring
Acronym: GLUCOSENS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GLUCOSENS
Record Dates: First submitted 2024-05-14; First posted 2024-06-25 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus; Hypoglycemia (Diabetic); Hypoglycemia Night; Hyperglycemia
Keywords: Blood glucose monitoring; point-of-care fingerstick capillary glucose monitoring; continuous glucose monitoring system; Patient satisfaction; Patient experience; Nursing staff's workload; Nursing staff's experience; accuracy
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia; Hyperglycemia; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: PERIOD 1: Point-of-care fingerstick glucose monitoring = Standard care, 110 patients
  * Substudy 1-3: 110 patients
  * Substudy 4: 14 patients of the 110 patients
  PERIOD 2: Point-of-care continuous glucose monitoring system = study Intervention 110 patients and 24 nursing staff
  * Substudy 1-3: 110 patients
  * Substudy 4: 20 patients of the 110 patients
  * Substudy 5*: 85 patients of the 110 patients
  * Substudy 6*: 85 patients of the 110 patients
  * Substudy 7: 24 nursing staff (20 surgical nursing staff and 4 specialized diabetes nurses)
  PERIOD 3*: Point-of-care fingerstick glucose monitoring = standard care + blinded sensor, 85 patients
  * Substudy 5*: 85 patients
  * Substudy 6*: 85 patients
    * Only conducted at Odense University Hospital
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- PERIOD 1: Point-of-care fingerstick glucose monitoring = standard care (No Intervention): Subjects' blood glucose levels are monitored using point-of-care fingerstick capillary glucose monitoring (standard care), which is conducted by surgical ward nurses according to a predefined schedule. Diabetes treatment management is overseen by specific in-house diabetes nurses. Treatment decisions are based on point-of-care fingerstick capillary glucose values.
- PERIOD 2: Glucose monitoring system as point-of-care = study intervention (Active Comparator): The sensor from the continuous glucose monitoring system is scanned by surgical nurses as point-of-care according to the predefined schedule, as in standard care. Monitoring is conducted by surgical ward nurses.
  Diabetes treatment management is overseen by specific in-house diabetes nurses. Diabetes nurses' treatment decisions are based on the continuous glucose monitoring system values.
  Interventions: Device: Abbott FreeStyle Libre System 2 Plus
- PERIOD 3: Point-of care fingerstick glucose monitoring = standard care + blinded sensor (Experimental): PERIOD 3: Same as for period 1, but with a blinded sensor (FreeStyle Libre Pro). The data from the blinded sensors are concealed from both participants and nurses and will be used for comparison with the experimental arm.
  This study period is only conducted at OUH.
  Interventions: Device: Abbott Freestyle Libre Pro

INTERVENTIONS:
Device: Abbott FreeStyle Libre System 2 Plus — The sensor is placed subcutaneously at the back of the participant's upper arm with one insertion and measures the subcutaneous glucose concentration.
  Arms: PERIOD 2: Glucose monitoring system as point-of-care = study intervention
Device: Abbott Freestyle Libre Pro — The sensor is placed subcutaneously at the back of the participant's upper arm with one insertion and measures the subcutaneous glucose concentration.
  Arms: PERIOD 3: Point-of care fingerstick glucose monitoring = standard care + blinded sensor

SUMMARY:
This clinical trial aims to compare a continuous glucose monitoring system with traditional fingerstick blood glucose monitoring. The study focuses on adult patients in general surgical wards who need regular blood glucose checks due to the risk of low or high blood sugar levels.

The goal is to learn if using a continuous glucose monitoring system is better than fingerstick monitoring in managing glucose levels, preventing complications, improving patient satisfaction and experience, reducing nursing staff workload, and improving nursing staff' experience. The study also compares the accuracy of glucose readings from the continuous glucose monitoring system with those from fingerstick tests and blood samples.

The hypothesis is that CGMS is accurate and effective for monitoring glucose levels in surgical patients. This could lead to better blood sugar control, fewer complications, shorter hospital stays, and improved experiences for both patients and nursing staff.

DETAILED DESCRIPTION:
Glucose control in surgical patients at risk of hyperglycemia and hypoglycemia is essential, as these conditions can lead to infections, poor surgical outcomes, prolonged hospital stays, and death. In 2022, the prevalence of diagnosed diabetes in Denmark was 6.2%. With the global incidence of diabetes on the rise, the number of patients requiring glucose control during surgical admissions is increasing.

Point-of-care (POC) fingerstick capillary glucose monitoring (FSGM) is standard in many hospitals; however, FSGM can be painful, disrupt sleep, and increase postoperative stress for patients. Additionally, it can be time-consuming, requiring up to two hours of nursing work per patient daily. This makes timely and prescribed glucose monitoring challenging in busy surgical wards, potentially leading to untreated hyperglycemia and hypoglycemia. Moreover, FSGM provides only a snapshot of glucose levels, without indicating whether glucose is stable, rising, or falling.

An alternative to FSGM is continuous glucose monitoring systems (CGMS), which measure glucose levels via a subcutaneous sensor every few minutes. CGMS is predominantly used in ambulatory settings and has been shown to improve glucose regulation. Several studies have confirmed the accuracy of CGMS compared to FSGM in surgical and medical wards, reporting an overall mean absolute relative difference ranging from 9.4 to 12.9, making it acceptable for use in surgical wards. Other studies have reported that CGMS in surgical and medical wards results in superior glycemic control, reduced hypoglycemia, insulin usage, and in-hospital complications, and detected significant duration of both hypo- and hyperglycemia despite protocolized perioperative diabetes management compared to FSGM.

Studies on patients' perspectives of CGMS have been limited to everyday life and outpatient settings. One review on patients with type 1 and 2 diabetes experienced improved convenience, control, and freedom by the use of CGMS but were also overwhelmed by data and frustrated by inaccuracy, and technical issues, which is consistent with findings from another review of patients with diabetes type 2. Another study reported that patients with type 2 diabetes found the technology helpful for disease management, although it could also serve as an unpleasant reminder of disease progression and cause discomfort.

One case report has described nurses' experiences with CGMS in hospital wards for patients with type 1 diabetes. The nurses experienced an increased workload due to difficulties hearing the device receiver, leading to more frequent patient observations.

In summary, CGMS has been reported to be safe and beneficial in ambulatory settings, while challenges and knowledge gaps remain in hospital wards. To date, no studies have compared glucose levels from CGMS with those from a laboratory plasma glucose analyzer as the reference. This study aims to investigate the effect of CGMS compared to FSGM in patients with hyperglycemia in general surgical wards on glucose levels, complications, length of hospital stay, and patient satisfaction and experience with glucose management during hospitalization and up to three months after discharge. Additionally, the study will investigate the nursing staff's workload and experience in the surgical ward, and the accuracy of CGMS throughout hospitalization, including during surgical procedures and medical imaging.

Seven substudies will be conducted:

Substudy 1 - Glucose levels and management for surgical patients in relation to hospitalization: Compares point-of-care glucose levels and management using point-of-care FSGM and point-of-care CGMS during hospitalization and FSGM and continuous glucose monitoring (CGM) up to three months after discharge.

Substudy 2 - Patient satisfaction with glucose monitoring and management in surgical wards: Compares patient satisfaction with glucose monitoring and management for surgical patients using point-of-care FSGM and point-of-care CGMS during hospitalization.

Substudy 3 - Nursing staff's glucose monitoring and management workload in the surgical ward: Compares the nursing staff's workload with point-of-care FSGM to point-of-care CGMS for surgical patients.

Substudy 4 (qualitative study) - Patient experience of glucose monitoring and management in relation to hospitalization in surgical wards: Compares the patient experience with point-of-care FSGM to point-of-care CGMS and glucose management during hospitalization in the surgical ward and one compares the patient experience of FSGM with CGM one month after discharge.

Substudy 5 - Continuous glucose level for surgical patients in relation to hospitalization in the surgical ward: Compares the continuous glucose levels when glucose monitoring and management are performed by point-of-care FSGM and point-of-care CGMS in the surgical ward. Further, it compares continuous glucose levels using point-of-care FSGM and CGM after discharge.

Substudy 6 - Accuracy of CGMS for surgical patients during hospitalization: Investigates the accuracy of CGMS by comparing CGMS data with FSGM and plasma glucose data.

Substudy 7 (qualitative study) - Nursing staff's experience with fingerstick monitoring and CGSM for surgical patients: Compares the nursing staff's experience with point-of-care FSGM to point-of-care CGMS and glucose management for surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients (≥ 18 years old) in surgical wards
* Glucose measurements at least 4 times (OUH) and 3 times (SUH) daily for at least three days, prescribed by surgeon
* Expected hospitalization for at least three days
* Communicates in Danish
* Signed a declaration of consent to study participation
* At risk of hypo- and hyperglycemia (with or without a diabetes diagnosis)
* Specific for substudy 4 inclusion criteria as above with the following add on: Patients being treated with insulin at discharge and patients residing within the OUH admission area.

Exclusion Criteria:

* Cognitively impaired patients
* Indication for glucose monitoring solely because of parenteral nutrition treatment
* Patients admitted with a CGMS
* Patients from the point-of-care fingerstick capillary glucose monitoring group cannot be included in the continuous glucose monitoring system group

Eligibility criteria solely for substudy 7

Inclusion Criteria:

* Nursing staff with at least one month of experience with both point-of-care fingerstick capillary glucose monitoring and continuous glucose monitoring system and are registered nurses or certified nursing assistants

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Substudy 1: Mean daytime and nocturnal point-of-care glucose levels | During hospitalization (up to 30 days)
  Point-of-care glucose levels measured by point-of-care continuous glucose monitoring system (CGMS) or point-of-care fingerstick capillary glucose monitoring (FSGM)
  Arm allocation:
  Period 1: FSGM Period 2: CGMS Number of measurements: minimum four times daily, hourly if fasting. Blood glucose measurement: mmol/L
Substudy 2: Patient-reported outcome on the convenience of glucose monitoring | During hospitalization (up to 30 days)
  Using the validated Danish version of the 22-item questionnaire: The Diabetes Treatment Satisfaction Questionnaire for Inpatients (DTSQ-IP), item 4: How convenient did you think the diabetes treatment was at hospitalization?
  Ranging from 0 - 6
  0 represents 'At no time' 6 represents 'At most of the time'
Substudy 3: Mean minutes surgical nursing staff spent on bedside glucose monitoring | During hospitalization (up to 30 days)
  Mean time: minutes.
  Data include:
  * Profession
  * Preparation (gathering materials, handwashing, disinfecting hands, putting on gloves, etc.)
  * Time for fingerstick or scanning of the continuous glucose monitor sensor
  * Display time of glucose level on device
  * Glucose level (mmol/L)
  * Actions taken after measurement (insulin injection, handwashing, documentation, disinfection, etc.)
  * Time for leaving the room
  * Time for completed procedure including documentation
  * Other observations made during the measurement
Substudy 5: Percentage of time in range (3.9-10.0 mmol/l) during the entire hospital stay | During hospitalization (up to 30 days)
  Percentage of time in range (3.9-10.0 mmol/l) during the entire hospital stay
Substudy 6: Differences in interstitial and plasma glucose | During hospitalization (up to 30 days)
  Glucose levels from CGMS are compared to plasma glucose, which are co-analyzed in blood tests.

SECONDARY OUTCOMES:
Substudy 1: • Mean dose of short-acting insulin (IE) | During hospitalization (up to 30 days)
  Unit: International units (IE)
Substudy 1: Mean dose of long-acting insulin (IE) | During hospitalization (up to 30 days)
  Unit: International units (IE)
eGFR | During hospitalization (up to 30 days)
  Estimated Glomerular Filtration Rate
Substudy 1: Complication: Sepsis | During hospitalization (up to 30 days)
  Defined as suspected or confirmed infection, as well as organ damage
Substudy 1: Complication: Acute kidney failure | During hospitalization (up to 30 days)
  Plasma creatinine, μmol/L
Substudy 1: Complication: First acute transfer to intensive care unit | During hospitalization (up to 30 days)
  The date for the first acute transfer to the intensive care unit and back to the surgical ward The number of days at the intensive care unit
  Unit: Days
Substudy 1: Complication: Second acute transfer to intensive care unit | During hospitalization (up to 30 days)
  The date for the second acute transfer to the intensive care unit and back to the surgical ward The number of days at the intensive care unit
  Unit: Days
Substudy 1: Complication: Infections | During hospitalization (up to 30 days)
  CRP, leucocytes, central body temperature. Unit: Days
Substudy 1: Complication: Antibiotics | During hospitalization (up to 30 days)
  Received antibiotics Unit: Days
Substudy 1: Complication: Bedsore | During hospitalization (up to 30 days)
  Presence of bedsore during hospitalization: yes/no
Substudy 1: Complication: Diabetes ketoacidosis | During hospitalization (up to 30 days)
  Diabetes ketoacidosis, defined as: pH < 7.30 and blood ketones > 3 mmol/L. Unit: Number of occurrence.
Substudy 1: Complication: Anastomotic leak | During hospitalization (up to 30 days)
  Presence of anastomotic leak during hospitalization: yes/no
Substudy 1: Readmission | 30-days after discharge from hospital
  Assesment of 30-day numbers of readmissions
Substudy 1: Mortality during hospitalization | During hospitalization (up to 30 days)
  Yes or no
Substudy 1: Mortality after discharge from hospital | 90-days after discharge from hospital
  Assesment of 90-day numbers of mortality.
Substudy 1: HbA1c three months after discharge | 90-days after discharge from hospital
  mmol/mol
Substudy 1: TIR and other established outcome derived from CGM | 90-days after discharge from hospital
  Percentage
Substudy 2: DTSQ-IP, treatment satisfaction (item 1) | During hospitalization (up to 30 days)
  Ranging from 0 - 6
  0 represents 'At no time' 6 represents 'Very satisfied'
Substudy 2: DTSQ-IP, experience with hyper- and hypoglycemia (items 2-3) | During hospitalization (up to 30 days)
  Ranging from 0 - 6
  0 represents 'At no time' 6 represents 'At most of the time'
Substudy 2: DTSQ-IP, treatment surveillance and flexibility (items 5+9), | During hospitalization (up to 30 days)
  Ranging from 0 - 6
  0 represents 'very unsatisfied"/"very inflexible' 6 represents ''very satisfied"very flexible"
Substudy 2: DTSQ-IP, treatment information, knowledge, and communication (items 15-18) | During hospitalization (up to 30 days)
  Ranging from 0 - 6
  0 represents 'very unsatisfied' 6 represents 'very satisfied'
Substudy 2: DTSQ-IP, contact with specialized diabetes nurses (items 20-21) | During hospitalization (up to 30 days)
  Ranging from 0 - 6
  0 represents 'very unsatisfied' 6 represents 'very satisfied'
Substudy 3: Mean minutes surgical nursing staff spent on reporting glucose levels and management to diabetes nurses | During hospitalization (up to 30 days)
  Measurement: Mean minutes
Substudy 3: Mean minutes the diabetes nurse spent in relation to the surgical patients | During hospitalization (up to 30 days)
  The mean minutes diabetes nurses spent collecting information about glucose levels and management, supervising patients and surgical professionals, and being supervised by endocrinologists.
Substudy 5: CGMS, time above range (TAR) 10,1-13.9 mmol/l | During hospitalization (up to 30 days)
  Percentage of time above range (TAR) 10,1-13.9 mmol/l
Substudy 5: CGMS, time above range (TAR) >13.9 mmol/l | During hospitalization (up to 30 days)
  Percentage of time above range >13.9 mmol/l
Substudy 5: CGMS, time below range 3.0-3.9 mmol/l | During hospitalization (up to 30 days)
  Percentage of time below range 3.0-3.9 mmol/l
Substudy 5: CGMS, time below range <3.0 | During hospitalization (up to 30 days)
  Percentage of time below range <3.0 mmol/l
Substudy 5: CGMS, standard deviation (SD) | During hospitalization (up to 30 days)
  mmol/l
Substudy 5: CGMS, coefficient of variation (CV) | During hospitalization (up to 30 days)
  SD divided by mean glucose level
Substudy 5: CGMS, mean glucose level daytime | During hospitalization (up to 30 days)
  mmol/l
Substudy 5: CGMS, mean glucose level night-time | During hospitalization (up to 30 days)
  mmol/l
Substudy 5: CGMS, Hypoglycemia level 1 (3.0-3.9 mmol/l) | During hospitalization (up to 30 days)
  Duration more than 15 consecutive minutes
Substudy 5: CGMS, hypoglycemia level 2 (<3.0 mmol/l) | During hospitalization (up to 30 days)
  Duration more than 15 consecutive minutes
Substudy 5: CGMS, number of hypoglycemic events in level 1 and 2, respectively | During hospitalization (up to 30 days)
  Number
Substudy 6: Differences in interstitial and capillary glucose | During hospitalization (up to 30 days)
  Glucose levels from CGMS are compared to FSGM data, which are co-analyzed in blood tests.

CONTACTS AND LOCATIONS:
Overall Officials: Karoline Schousboe, MD, PhD, Study Chair — Steno Diabetes Center Odense, Odense University Hospital; Helen Schultz, RN, PhD, Study Chair — The Department of Surgery, Odense University Hospital
Locations (2):
- Denmark (2):
  - Department of Surgery, Zealand University Hospital, Køge, Køge
  - The Department of Surgery, Odense Univeristy Hospital, Odense, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berrios-Torres SI, Umscheid CA, Bratzler DW, Leas B, Stone EC, Kelz RR, Reinke CE, Morgan S, Solomkin JS, Mazuski JE, Dellinger EP, Itani KMF, Berbari EF, Segreti J, Parvizi J, Blanchard J, Allen G, Kluytmans JAJW, Donlan R, Schecter WP; Healthcare Infection Control Practices Advisory Committee. Centers for Disease Control and Prevention Guideline for the Prevention of Surgical Site Infection, 2017. JAMA Surg. 2017 Aug 1;152(8):784-791. doi: 10.1001/jamasurg.2017.0904. PMID 28467526
- [Background] Kotagal M, Symons RG, Hirsch IB, Umpierrez GE, Dellinger EP, Farrokhi ET, Flum DR; SCOAP-CERTAIN Collaborative. Perioperative hyperglycemia and risk of adverse events among patients with and without diabetes. Ann Surg. 2015 Jan;261(1):97-103. doi: 10.1097/SLA.0000000000000688. PMID 25133932
- [Background] Carstensen B, Ronn PF, Jorgensen ME. Prevalence, incidence and mortality of type 1 and type 2 diabetes in Denmark 1996-2016. BMJ Open Diabetes Res Care. 2020 May;8(1):e001071. doi: 10.1136/bmjdrc-2019-001071. PMID 32475839
- [Background] Carstensen B, Ronn PF, Jorgensen ME. Components of diabetes prevalence in Denmark 1996-2016 and future trends until 2030. BMJ Open Diabetes Res Care. 2020 Aug;8(1):e001064. doi: 10.1136/bmjdrc-2019-001064. PMID 32784246
- [Background] Stahl-Pehe A, Kamrath C, Prinz N, Kapellen T, Menzel U, Kordonouri O, Schwab KO, Bechtold-Dalla Pozza S, Rosenbauer J, Holl RW. Prevalence of type 1 and type 2 diabetes in children and adolescents in Germany from 2002 to 2020: A study based on electronic health record data from the DPV registry. J Diabetes. 2022 Dec;14(12):840-850. doi: 10.1111/1753-0407.13339. Epub 2022 Dec 14. PMID 36515004
- [Background] Galindo RJ, Migdal AL, Davis GM, Urrutia MA, Albury B, Zambrano C, Vellanki P, Pasquel FJ, Fayfman M, Peng L, Umpierrez GE. Comparison of the FreeStyle Libre Pro Flash Continuous Glucose Monitoring (CGM) System and Point-of-Care Capillary Glucose Testing in Hospitalized Patients With Type 2 Diabetes Treated With Basal-Bolus Insulin Regimen. Diabetes Care. 2020 Nov;43(11):2730-2735. doi: 10.2337/dc19-2073. Epub 2020 Jul 8. PMID 32641372
- [Background] American Diabetes Association Professional Practice Committee. 16. Diabetes Care in the Hospital: Standards of Medical Care in Diabetes-2022. Diabetes Care. 2022 Jan 1;45(Suppl 1):S244-S253. doi: 10.2337/dc22-S016. PMID 34964884
- [Background] Mianowska B, Mlynarski W, Szadkowska I, Szadkowska A. Evaluation of Three Lancing Devices: What Do Blood Volume and Lancing Pain Depend On? J Diabetes Sci Technol. 2021 Sep;15(5):1076-1083. doi: 10.1177/1932296820949930. Epub 2020 Aug 17. PMID 32856497
- [Background] Kocher S, Tshiananga JK, Koubek R. Comparison of lancing devices for self-monitoring of blood glucose regarding lancing pain. J Diabetes Sci Technol. 2009 Sep 1;3(5):1136-43. doi: 10.1177/193229680900300517. PMID 20144427
- [Background] Aragon D. Evaluation of nursing work effort and perceptions about blood glucose testing in tight glycemic control. Am J Crit Care. 2006 Jul;15(4):370-7. PMID 16823014
- [Background] Gothong C, Singh LG, Satyarengga M, Spanakis EK. Continuous glucose monitoring in the hospital: an update in the era of COVID-19. Curr Opin Endocrinol Diabetes Obes. 2022 Feb 1;29(1):1-9. doi: 10.1097/MED.0000000000000693. PMID 34845159
- [Background] Lin R, Brown F, James S, Jones J, Ekinci E. Continuous glucose monitoring: A review of the evidence in type 1 and 2 diabetes mellitus. Diabet Med. 2021 May;38(5):e14528. doi: 10.1111/dme.14528. Epub 2021 Mar 6. PMID 33496979
- [Background] Carlsson CJ, Norgaard K, Oxboll AB, Sogaard MIV, Achiam MP, Jorgensen LN, Eiberg JP, Palm H, Sorensen HBD, Meyhof CS, Aasvang EK. Continuous Glucose Monitoring Reveals Perioperative Hypoglycemia in Most Patients With Diabetes Undergoing Major Surgery: A Prospective Cohort Study. Ann Surg. 2023 Apr 1;277(4):603-611. doi: 10.1097/SLA.0000000000005246. Epub 2021 Oct 8. PMID 35129526
- [Background] Cavalcante Lima Chagas G, Teixeira L, R C Clemente M, Cavalcante Lima Chagas R, Santinelli Pestana DV, Rodrigues Silva Sombra L, B Lima B, J Galindo R, Abreu M. Use of continuous glucose monitoring and point-of-care glucose testing in hospitalized patients with diabetes mellitus in non-intensive care unit settings: A systematic review and meta-analysis of randomized controlled trials. Diabetes Res Clin Pract. 2025 Feb;220:111986. doi: 10.1016/j.diabres.2024.111986. Epub 2025 Jan 9. PMID 39798897
- [Background] Olsen MT, Klarskov CK, Jensen SH, Rasmussen LM, Lindegaard B, Andersen JA, Gottlieb H, Lunding S, Pedersen-Bjergaard U, Hansen KB, Kristensen PL. In-Hospital Diabetes Management by a Diabetes Team and Insulin Titration Algorithms Based on Continuous Glucose Monitoring or Point-of-Care Glucose Testing in Patients With Type 2 Diabetes (DIATEC): A Randomized Controlled Trial. Diabetes Care. 2025 Apr 1;48(4):569-578. doi: 10.2337/dc24-2222. PMID 39887698
- [Background] Natale P, Chen S, Chow CK, Cheung NW, Martinez-Martin D, Caillaud C, Scholes-Robertson N, Kelly A, Craig JC, Strippoli G, Jaure A. Patient experiences of continuous glucose monitoring and sensor-augmented insulin pump therapy for diabetes: A systematic review of qualitative studies. J Diabetes. 2023 Dec;15(12):1048-1069. doi: 10.1111/1753-0407.13454. Epub 2023 Aug 8. PMID 37551735
- [Background] Taylor PJ, Thompson CH, Brinkworth GD. Effectiveness and acceptability of continuous glucose monitoring for type 2 diabetes management: A narrative review. J Diabetes Investig. 2018 Jul;9(4):713-725. doi: 10.1111/jdi.12807. Epub 2018 Mar 1. PMID 29380542
- [Background] Chiu CJ, Chou YH, Chen YJ, Du YF. Impact of New Technologies for Middle-Aged and Older Patients: In-Depth Interviews With Type 2 Diabetes Patients Using Continuous Glucose Monitoring. JMIR Diabetes. 2019 Feb 21;4(1):e10992. doi: 10.2196/10992. PMID 30789351
- [Background] Wang M, Singh LG, Spanakis EK. Advancing the Use of CGM Devices in a Non-ICU Setting. J Diabetes Sci Technol. 2019 Jul;13(4):674-681. doi: 10.1177/1932296818821094. Epub 2019 Jan 13. PMID 30636449
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Spanakis EK, Cook CB, Kulasa K, Aloi JA, Bally L, Davis G, Dungan KM, Galindo RJ, Mendez CE, Pasquel FJ, Shah VN, Umpierrez GE, Aaron RE, Tian T, Yeung AM, Huang J, Klonoff DC. A Consensus Statement for Continuous Glucose Monitoring Metrics for Inpatient Clinical Trials. J Diabetes Sci Technol. 2023 Nov;17(6):1527-1552. doi: 10.1177/19322968231191104. Epub 2023 Aug 17. PMID 37592726
- [Background] Rutter CL, Jones C, Dhatariya KK, James J, Irvine L, Wilson EC, Singh H, Walden E, Holland R, Harvey I, Bradley C, Sampson MJ. Determining in-patient diabetes treatment satisfaction in the UK--the DIPSat study. Diabet Med. 2013 Jun;30(6):731-8. doi: 10.1111/dme.12095. Epub 2013 Mar 6. PMID 23350704
- [Background] Sampson MJ, Singh H, Dhatariya KK, Jones C, Walden E, Bradley C. Psychometric validation and use of a novel diabetes in-patient treatment satisfaction questionnaire. Diabet Med. 2009 Jul;26(7):729-35. doi: 10.1111/j.1464-5491.2009.02754.x. PMID 19573123
- [Background] Verissimo D, Vinhais J, Ivo C, Martins AC, Nunes E Silva J, Passos D, Lopes L, Jacome de Castro J, Marcelino M. Continuous Glucose Monitoring vs. Capillary Blood Glucose in Hospitalized Type 2 Diabetes Patients. Cureus. 2023 Aug 21;15(8):e43832. doi: 10.7759/cureus.43832. eCollection 2023 Aug. PMID 37736430
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Derived] Schultz H, Petersen MC, Nielsen KB, Abrahamsen L, Nielsen TD, Joergensen UL, Thomsen TL, Schousboe K. GLUCOSENS study protocol: a continuous glucose monitoring system compared to fingerstick glucose monitoring in surgical wards - a two-centre before-after clinical trial. BMJ Open. 2025 Apr 2;15(4):e095503. doi: 10.1136/bmjopen-2024-095503. PMID 40180373
- See also: Prevalence of patients with diagnosed diabetes in Denmark in 2022 — https://diabetes.dk/forskning/viden-om-diabetes/diabetes-i-danmark
- See also: Incidence of diabetes worldwide — https://www.who.int/health-topics/diabetes?gad_source=1&gclid=EAIaIQobChMIv8fij6DnhQMVS0CRBR3--Q_yEAAYASAAEgLq_vD_BwE#tab=tab_1
- See also: User's guide for Abbotts' freestyle libre devices — https://www.diabetescare.abbott/support/manuals/dk.html